CLINICAL TRIAL: NCT05300594
Title: Double-blind Randomized Control Trial Versus Placebo to Assess the Daily Consumption Audistim® Day/Night on Hearing Comfort and Quality of Life of Patients With Chronic Tinnitus
Brief Title: Effect of Audistim® Day/Night on Hearing Comfort and Patient Quality of Life of Patients With Chronic Tinnitus.
Acronym: TINNITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEN Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: C1694
Record Dates: First submitted 2022-03-15; First posted 2022-03-29 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-08

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Plant Extracts; Vitamins; Minerals

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audistim (Experimental): The participants ingest the experimental product every day for 3 months. The experimental product contains a combination of plant extracts, vitamins and trace elements presented in 2 formulas: a day tablet (to be swallowed in the morning) and a night tablet (to be swallowed in the evening before going to bed).
  Interventions: Dietary Supplement: Plant extracts, vitamins and mineral
- Placebo (Placebo Comparator): Participants ingest the placebo product every day for 3 months .The placebo is strictly identical in appearance to the experimental product and contains only excipients.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Plant extracts, vitamins and mineral — Day tablet every day during 3 months : Magnesium (75 mg), Ginkgo Biloba extract (40 mg), hawthorn extract (37,5 mg), L-Theanin (50 mg) , Niacin (16mg), Quercetin (25mg), B12 Vitamin (2,5 µg), B6 Vitamin (1,4 mg), Thiamin (1,1 mg)
  Night tablet every evening during 3 months : Magnesium (37,5 mg), Ginkgo Biloba extract (40 mg), Eschscholzia californica extract (40 mg), Zinc (10 mg), Melatonin (1mg), Lemon balm extract (80 mg), Tryptocetyn (65 mg)
  Other Names: Audistim Day Night
  Arms: Audistim
Dietary Supplement: Placebo — Day tablet every morning during 3 months : Excipients; Night tablet every evening during 3 months : Excipients
  Arms: Placebo

SUMMARY:
Tinnitus is a widespread problem that affects the quality of life of millions globally.

Few treatments have been found to be effective for subjective tinnitus and to have a significant improvement on quality of life. In subjective tinnitus, neither an external nor endogenous sound source is present; instead, the tinnitus is caused by abnormal bioelectric, biomechanical, or biochemical activity in the inner ear and/or central nervous system.

The precise role of the numerous extra-auditory structures that contribute to the pathophysiology of tinnitus is difficult to establish. Some of them participate in the creation or in the chronification of tinnitus and some in the psychological reactions to the tinnitus.

Audistim contains ingredients with a specific composition based upon the multifactorial causal theory; which involves auditory, attentional, memory, and emotional systems. These different systems are being targeted by the ingredients and their specific proportioning. Also the antioxidant theory is involved in the creation of Audistim, it states that the reactive oxygen species play an important microcirculatory role in the pathology of the inner ear and the peripheral and central pathways. These components help to treat the multitude of causing factors and in that way improve the quality of life.

DETAILED DESCRIPTION:
Participants are allocated in test (dietary supplement) or placebo group according a ratio 1:1.

The participants are asked to consume daily the investigational product for 3 months. The effect of the dietary supplement is assessed by comparing chronic tinnitus evolvement between groups.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from subjective tinnitus for at least 6 months;
* Tinnitus whose level of severity is defined by THI values ≥12 and ≤ 76;
* Having given their written and informed consent to participate in the study.

Main Exclusion Criteria:

* Severe Tinnitus (grade 5 corresponding to a THI ≥78);
* Tinnitus with no or very slight impact on daily life (<2 out of a 10-point numerical scale);
* Unilateral or bilateral cophosis;
* Holder of an implant (cochlear, bone anchor);
* Wearer of an airborne hearing aid for less than 6 months;
* Suffering from hearing pathologies (Menière's disease, chronic otitis, vestibular neuritis, neuroma, otosclerosis cholesteatoma);
* With otitis, earwax plug or damage to the eardrum inclusion;
* Having started treatment with ototoxic drugs (anti-inflammatory, anti-coagulant, anti-arrhythmic, hypotensive, anti- depressants, MAOIs, Benzodiazepines, opioids) in the past 2 months;
* Pharmacological treatment of tinnitus during the last 2 months;
* Non-pharmacological treatments for tinnitus in the last 2 months: cognitive-behavioral therapy, habituation treatments or other therapies;
* Taking food supplements containing one of the compounds of the product under study in the last month;
* Known allergy to one of the compounds of the product under study;
* Suffering from heart disease, hypertension, diabetes, autoimmune disease, inflammatory disease or pathology major or progressive;
* Epileptic subject.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline Tinnitus Handicap Inventory (THI) score to 3 months | at month 0 (at inclusion), at month 3 (after 3 months of supplementation)
  THI is a widely used questionnaire to assess the severity of tinnitus. It is composed of 25 items in total, with functional (11 items), emotional (9 items), and catastrophic (5 items) subscales. Three response options (0=none, 2=sometimes, 4=always) are available for each item, and the total score is calculated by summing all responses. A total possible score of THI ranges from 0 to 100, and the higher score of THI represents greater handicap from tinnitus. The THI score of 0-16 means "no or slight handicap", 18 to 36 indicates "mild", 38 to 56 indicates "moderate", 58 to 76 indicates "severe", and a score of 78-100 is classified as "catastrophic handicap".

SECONDARY OUTCOMES:
Change from baseline Tinnitus Handicap Inventory (THI) score to 1 month | at month 0 (at inclusion), at month 1 (after one month of supplementation)
  THI is a widely used questionnaire to assess the severity of tinnitus. It is composed of 25 items in total, with functional (11 items), emotional (9 items), and catastrophic (5 items) subscales. Three response options (0=none, 2=sometimes, 4=always) are available for each item, and the total score is calculated by summing all responses. A total possible score of THI ranges from 0 to 100, and the higher score of THI represents greater handicap from tinnitus. The THI score of 0-16 means "no or slight handicap", 18 to 36 indicates "mild", 38 to 56 indicates "moderate", 58 to 76 indicates "severe", and a score of 78-100 is classified as "catastrophic handicap".
Psycological Stress Measure scale (MSP-9) | at month 0 (at inclusion), at month 1 (after one month of supplementation), at month 3 (after 3 months of supplementation)
  The scale, no matter how many items it contains, is composed of symptom-descriptors of affective, cognitive, behavioral and physical problems. The respondent indicates to what extent the items describe him for the last 4 or 5 days. Examples of items (from the 53-item version): "1- I am tense or tense, 2- I feel my throat tight or I have a dry mouth, 3- I take more two alcohol drinks a day". Response options range from 1 (=not at all) to 8 (=extremely).The authors argue that the 9-item version displays the same psychometric qualities of reliability and internal consistency (0.89) as the 49- and 25-item versions.
Pittsburgh sleep quality index | at month 0 (at inclusion), at month 1 (after one month of supplementation), at month 3 (after 3 months of supplementation)
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval.Consisting of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Patient Global Impression of Improvement (PGII) | at month 1 (after one month of supplementation), at month 3 (after 3 months of supplementation)
  The Patient Global Imression of Improvement (PGI-I) is a 7 point scale that requires the patient to assess himself how his illness has improved or worsened relative to a baseline state at the beginning of the intervention. "Compared to your condition at baseline, your condition has...?" and rated as:
  Very much improved Much improved Minimally improved No change Minimally worse Much worse Very much worse
Clinical Global Impression of Improvement (CGI-I) | at month 1 (after one month of supplementation), at month 3 (after 3 months of supplementation)
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention."Compared to the patient's condition at baseline, this patient's [average] condition has...?" and rated as:
  Very much improved Much improved Minimally improved No change Minimally worse Much worse Very much worse

CONTACTS AND LOCATIONS:
Locations (1):
- CEN Nutriment, Dijon, Bourgogne-Franche-Comté, France